CLINICAL TRIAL: NCT03942887
Title: Evaluating Clinical and Immunological Effects of Rituximab With Cyclophosphamide Compared to Rituximab Alone in AAV Patients
Brief Title: Exploring Durable Remission With Rituximab in Antineutrophil Cytoplasmic Antibody(ANCA)-Associated Vasculitis
Acronym: ENDURRANCE-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Y.K.Onno Teng, Nephrologist, head of outpatient clinic nephrology department, drs. Y.K.O. Teng, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL67515.058.18
Record Dates: First submitted 2019-04-08; First posted 2019-05-08 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: ANCA Associated Vasculitis
Keywords: ANCA; Crescentic glomerulonephritis; systemic autoimmune disease; Renal failure; Renal insufficiency; small vessel vasculitis; GPA; MPA
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Renal Insufficiency | interventions — Rituximab; Cyclophosphamide; Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: open-label, 1:1 randomized, prospective study between RTX with cyclophosphamide and RTX alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Active Comparator): Patients will be intravenously treated with Rituximab 1000mg (or biosimilar) in the first week and receive a 2nd dosage of 1000mg 14 days later. Before every infusion of Rituximab patients will receive intravenous methylprednisolone 100mg together with oral acetaminophen 1000 mg and and intravenous Tavegil 2 mg.
  Interventions: Drug: Rituximab; Drug: Methylprednisolone; Drug: Prednisolone
- Rituximab plus low-dose cyclophosphamide (Active Comparator): 5.1.2. Cyclophosphamide Patients will be intravenously treated with a total of 6 infusions of cyclophosphamide 500mg every 2 weeks. Before every infusion of cyclophosphamide patients will receive intravenous granisetron to prevent nausea.
  Interventions: Drug: Rituximab; Drug: endoxan; Drug: Methylprednisolone; Drug: Prednisolone

INTERVENTIONS:
Drug: Rituximab — Patients will be intravenously treated with Rituximab 1000mg (or biosimilar) in the first week and receive a 2nd dosage of 1000mg 14 days later. Before every infusion of Rituximab patients will receive intravenous methylprednisolone 100mg together with oral acetaminophen 1000 mg and and intravenous Tavegil 2 mg. At any time during the study, a rituximab biosimilar is allowed as a substitute for the bio-originator rituximab.
  Other Names: anti-cd20
Drug: endoxan — Patients will be intravenously treated with a total of 6 infusions of cyclophosphamide 500mg every 2 weeks. Before every infusion of cyclophosphamide patients will receive intravenous granisetron to prevent nausea.
  Other Names: cyclophosphamide
  Arms: Rituximab plus low-dose cyclophosphamide
Drug: Methylprednisolone — Patients are given 1-3 pulses of 500mg methylprednisolone i.v. up to a maximum cumulative dose of 3000mg, taking into account any doses of intravenous methylprednisolone administered within 12 weeks prior to screening.
  Other Names: solumedrol
Drug: Prednisolone — after intravenous pulse methylprednisolone, oral prednisolone will be given at a dose of 1mg/kg daily and tapered according to the recommendations
  Other Names: corticosteroid

SUMMARY:
Most recent insights in the treatment for patients with ANCA-associated vasculitis (AAV) have demonstrated that 'tailored' maintenance treatment with rituximab (RTX) is effective to achieve durable remission of disease. As such, RTX re-treatment can be tailored on the basis of relevant clinical and immunological parameters in AAV patients. Now, the present study intends to evaluate whether combining rituximab with cyclophosphamide is superior to current standard of care with rituximab only to induce a favorable clinical and immunological state in AAV patients and can thereby reduce the number of tailored re-treatments with rituximab.

DETAILED DESCRIPTION:
Objectives: The primary objective is to prove that the combination of RTX and low-dose CYC reduces the number of RTX infusions needed to maintain clinical remission over 2 years. The secondary objectives are measurements for minimal residual auto-immunity (MRA) such as time to ANCA seronegativity, proportion of seronegativity, time to ANCA return, proportion of ANCA return, duration of B-cell depletion and the composition of the memory B-cell and plasma cell populations. Other secondary objectives are the potential association between MRA and disease flares, and the evaluation of (severe) adverse events, cost-effectiveness and quality of life Study design: open-label, multicenter, 1:1 randomized, prospective study Study population: Adult AAV patients with a clinical diagnosis of granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA) who have 'generalised disease' and a positive ANCA-test for anti-PR3 or anti-MPO.

Intervention: In addition to standard of care corticosteroid therapy, AAV patients will be randomized to receive either standard induction therapy with 2 infusions of RTX 1000 mg or induction therapy combining 2 infusions of RTX 1000 mg with 6 infusions of low dose intravenous cyclophosphamide 500mg. Thereafter, as part of standard of care patients will receive tailored RTX re-treatment as maintenance therapy.

Main study parameters: AAV patients will be evaluated for the cumulative number of events for tailored RTX retreatments needed to maintain clinical remission over 2 years. Also, AAV patients will be evaluated for MRA by prospectively and consecutively studying ANCA levels and B-cell depletion by standard flowcytometry at predefined timepoints. Additionally, the study will perform safety and toxicity monitoring according to WHO toxicity criteria and evaluate the clinical response, the number of moderate and severe flares during study follow-up, the cost-effectiveness, and the quality of life of patients.

Study duration: 2 years

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the study must meet the following inclusion criteria:

1. Clinical diagnosis of granulomatosis with polyangiitis (GPA) or microscopic Polyangiitis (MPA), consistent with Chapel-Hill Consensus Conference definitions26
2. Aged at least 18 years, with newly-diagnosed or relapsed AAV with 'generalised disease', defined as involvement of at least one major organ (e.g. kidney, lung, heart, peripheral or central nervous system), requiring induction treatment with cyclophosphamide or rituximab
3. Positive test for anti-PR3 or anti-MPO (current or historic)
4. Willing and able to give written Informed Consent and to comply with the requirements of the study protocol

Exclusion criteria:

Subjects will be excluded from participation if they meet any of the following exclusion criteria:

1. Pregnant or breast-feeding
2. Active pregnancy, as proven by a positive urine beta-HCG test or a positive serum beta-HCG
3. Significant hypogammaglobulinemia (IgG < 4.0 g/L) or an IgA deficiency (IgA < 0.1 g/L)
4. Active infection not compatible with start of remission-induction therapy in the opinion of the treating physician and/or investigator, e.g.:

   * Serological evidence of viral hepatitis defined as: patients positive for HbsAg test or HBcAb or a positive hepatitis C antibody not treated with antiviral medication
   * Have a historically positive HIV test or test positive at screening for HIV
5. Have a history of a primary immunodeficiency
6. Have a significant infection history that in the opinion of the investigator would make the candidate unsuitable for the study
7. Have a neutrophil count of < 1.5x10E9/L
8. Evidence of hepatic disease: AST, ALT, alkaline phosphatase, or bilirubin > 3 times the upper limit of normal before start of dosing
9. Have any other clinically significant abnormal laboratory value in the opinion of the investigator
10. Required dialysis or plasma exchange within 12 weeks prior to screening
11. Received intravenous glucocorticoids, >3000mg methylprednisolone equivalent, within 4 weeks prior to screening
12. Immunization with a live vaccine 1 month before screening
13. History or presence of any medical condition or disease which, in the opinion of the Investigator, may place the patient at unacceptable risk for study participation.
14. Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of tailored RTX infusions | 2 years
  The primary outcome is the number of RTX infusions needed to maintain clinical remission over 2 years

SECONDARY OUTCOMES:
Time | 2 years
  - time to a ANCA negative test
ANCA reappearance | 2 years
  - Percentage of patients that have ANCA return during follow-up
B cell depletion | 2 years
  - duration of B-cell depletion
Remission and relaps rate | 2 years
  - to compare disease controle between arms
Number of adverse events | 2 years
  - to assess the safety parameters of each treatment arm including adverse events according to WHO toxicity criteria, time to immune reconstitution and recording of infectious events
Quality of Life by AAV-PRO | 2 years
  assess quality of life by AAV-PRO
BVAS | 2 years
  Disease activity will be assessed by BVAS
concomitant immunosuppressants | 2 years
  Disease activity assessed by (the reduction of) concomitant immunosuppressants
Kidney function | 2 years
  Return of kidney function will be assessed.
Biomarker for inflammation | 2 years
  Disease activity assessed by ESR

CONTACTS AND LOCATIONS:
Overall Officials: YKO Teng, MD, PhD, Principal Investigator — LUMC Leiden
Locations (4):
- Netherlands (4):
  - Leiden University Medical Center, Leiden, South Holland
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Meander Medical Center, Amersfoort
  - HagaZiekenhuis, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dirikgil E, van Leeuwen JR, Bredewold OW, Ray A, Jonker JT, Soonawala D, Remmelts HHF, van Dam B, Bos WJ, van Kooten C, Rotmans J, Rabelink T, Teng YKO. ExploriNg DUrable Remission with Rituximab in ANCA-associatEd vasculitis (ENDURRANCE trial): protocol for a randomised controlled trial. BMJ Open. 2022 Sep 21;12(9):e061339. doi: 10.1136/bmjopen-2022-061339. PMID 36130755